CLINICAL TRIAL: NCT04846673
Title: Efficacy and Safety of Pregabalin and Alpha-lipoic Acid Combination Versus Each Monotherapy in Patients With Diabetic Peripheral Neuropathy: a Randomized, Parallel, Open-label, Multicenter, Phase IV Clinical Trial (OPTIMUM Trial)
Brief Title: Pregabalin and Alpha-lipoic Acid Combination Versus Each Monotherapy in Patients With Diabetic Peripheral Neuropathy
Acronym: OPTIMUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC045
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Pregabalin; Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pregabalin and alpha-lipoic acid combination therapy (Experimental): Alpha-lipoic acid 480 mg/tablet once daily before breakfast and Pregabalin 150 mg/tablet once daily before bedtime will be administrated for 12 weeks.
  Interventions: Drug: Pregabalin 150mg + Alpha-lipoic acid 480mg
- Pregabalin monotherapy (Experimental): Pregabalin 150 mg/tablet once daily before bedtime will be administrated for 12 weeks.
  Interventions: Drug: Pregabalin 150mg
- Alpha-lipoic acid monotherapy (Active Comparator): Alpha-lipoic acid 480 mg/tablet once daily before breakfast will be administrated for 12 weeks.
  Interventions: Drug: Alpha-Lipoic Acid 480mg

INTERVENTIONS:
Drug: Pregabalin 150mg + Alpha-lipoic acid 480mg — Pregabalin qd + alpha-lipoic acid qd
  Arms: Pregabalin and alpha-lipoic acid combination therapy
Drug: Pregabalin 150mg — pregabalin qd
  Arms: Pregabalin monotherapy
Drug: Alpha-Lipoic Acid 480mg — alpha-lipoic acid qd
  Arms: Alpha-lipoic acid monotherapy

SUMMARY:
This study is a randomized, parallel, open-label, multicenter, phase IV clinical trial to assess the efficacy and safety of pregabalin and alpha-lipoic acid combination compared with each monotherapy in patients with diabetic peripheral neuropathy for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 19 to 75
* type 2 diabetes mellitus with HbA1c (Hemoglobin A1c) ≤ 10 %
* peripheral (eg. hands, feet) neuropathic pain (eg. abnormal sensations, numbness, pain, etc.) within 3 months (12 weeks)
* diagnosed with diabetic peripheral neuropathy (DPN)
* VAS pain score ≥ 40 mm
* written informed consent

Exclusion Criteria:

* brittle diabetes mellitus
* ALT (Alanine Transaminase), AST (Aspartate Transaminase), CPK (Creatine Phosphokinase) level ≥ 3 times the upper limit of normal (UNL) or active liver disease
* severe renal impairment (eGFR (estimated glomerular filtration rate) < 60 mL/min/ 1.73m2)
* treated with antiepileptic drugs within 1 week at randomization
* other nervous system or neuropathic disorders that may affect pain evaluation
* oral drug administration is not possible, or hypersensitive or allergic to pregabalin, r-thioctic acid tromethamine, thioctic acid, and other excipients
* pregnant, lactating, or childbearing potential
* alcoholics, drug abusers, and patients who are difficult to participate in clinical trials due to psychological and emotional problems
* have participated in other clinical trials within 30 days at screening

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | 12 weeks

SECONDARY OUTCOMES:
visual analogue scale (VAS) | 6 weeks
visual analogue scale (VAS) reduction rate of more than 30% | 6 weeks, 12 weeks
visual analogue scale (VAS) reduction rate of more than 50% | 6 weeks, 12 weeks
brief pain inventory Korean version, BPI-K | 6 weeks, 12 weeks
total symptom score, TSS | 6 weeks, 12 weeks
pain detect questionnaire, PD-Q | 6 weeks, 12 weeks
3 level version of Euro-Qol-5 dimensions, EQ-5D-3L | 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jongchul Won, Principal Investigator — Inje University
Locations (14):
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Chosun University Hospital, School of Medicine, Chosun University, Gwangju
  - Dongtan Sacred Heart Hospital, Hallym University College of Medicine, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - The Catholic University of Korea, Incheon ST. Mary's Hospital, Incheon
  - Jeju National University College of Medicine, Jeju City
  - Jeonbuk National University Hospital, Jeollabuk-do
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul St.Mary's Hospital, The Catholic University of Korea, Seoul
  - Yeouido St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Ulsan University Hospital, College of Medicine University of Ulsan, Ulsan